CLINICAL TRIAL: NCT01267721
Title: Macrophage Migration Inhibitory Factor (MIF) as a Marker of Perioperative Inflammatory Reaction During Heart Surgery
Brief Title: Macrophage Migration Inhibitory Factor (MIF)- Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: CTC-A10-029
Record Dates: First submitted 2010-12-22; First posted 2010-12-28 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Heart Surgery
Keywords: heart surgery
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — inflammatory markers (different)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: A single group of 100 consecutive patients will undergo additional blood sampling at different time points
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling at various time points. Additional 92 mL blood.

SUMMARY:
It has been repeatedly demonstrated that cardiac surgery with the use of extracorporeal circulation elicits a systemic inflammatory response and provokes ischemia-reperfusion related oxidative stress which could further lead to the development of organ failure in critically ill patients. Perioperative levels of macrophage migration inhibitory factor (MIF) and other inflammatory mediators could be involved in adverse outcomes in cardiac surgery.

DETAILED DESCRIPTION:
The trace element selenium (Se) serves as an essential co-factor for the antioxidant enzymes Thioredoxin - reductase (TRR) and many other antioxidant enzymes, which protect tissues from oxidative stress. In septic patients it has previously been shown that thioredoxin, a TRR regulated Redox Enzyme, has the ability to suppress the synthesis of MIF.

Aim of the present study is therefore to investigate the relation between perioperative selenium decrease and the reduction of TRR activity with a possible release of MIF during the inflammatory response after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years of age
* open heart surgery and use of heart-lung-device
* informed consent has been obtained

Exclusion Criteria:

* under 18 years of age
* emergency cases
* informed consent cannot be obtained
* pregnancy or patient is breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open heart surgery and use of heart lung device
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pilot study: correlation between clinical and lab parameters | two months
  To assess the importance of the MIF ligand/receptor family in a large cohort of patients (n=100) undergoing cardiac surgery and to characterize the underlying molecular events.
  Possible correlation between several clinical and laboratory parameters will be analyzed. This is a pilot study to generate hints at future items to be studied in controlled trials.

SECONDARY OUTCOMES:
Secondary Outcome | two months
  * Correlation between perioperative MIF and MIF-2 levels and postoperative outcome
  * Measurement of sCD74/MIF complex
  * Determination of MIF polymorphism and its significance on clinical outcome
  * perioperative inflammation
  * organ injury

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Rex, PD Dr. med., Principal Investigator — RWTH Aachen University Hospital
Locations (1):
- RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia, Germany